CLINICAL TRIAL: NCT00002131
Title: A Pilot Study of OPC-8212 (Vesnarinone) in Persons With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka America Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 234D; 22-93-254
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antiviral Agents; vesnarinone
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — vesnarinone

INTERVENTIONS:
Drug: Vesnarinone

SUMMARY:
To examine the safety and efficacy of two doses of vesnarinone in patients with AIDS-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
Twenty-eight patients (14 per cohort) receive daily vesnarinone at one of two doses. At least seven patients at the lower dose must have completed 2 weeks of therapy before subsequent patients are entered at the higher dose. Patients who successfully complete 16 weeks of treatment may receive maintenance therapy for the duration of the study (approximately 12-18 months).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii, candida, and mycobacteria.
* Acyclovir as acute treatment for herpes outbreaks.

Concurrent Treatment:

Allowed:

* Limited electron-beam radiation therapy to non-marker lesions for treatment of Kaposi's sarcoma.

Patients must have:

* Documented HIV infection.
* Kaposi's sarcoma.
* No current constitutional signs of HIV disease or AIDS-defining conditions other than Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active malignancy other than Kaposi's sarcoma, cutaneous basal cell carcinoma, or in situ carcinoma of the cervix.
* Current significant cardiac disease or anomaly (including prolonged QTC on EKG).
* Abnormal cardio-thoracic ratio on chest x-ray.

Concurrent Medication:

Excluded:

* Antiretroviral agents, including ddI, ddC, AZT, and d4T.
* Immunosuppressive agents.
* Investigational HIV drugs/therapies including vaccines (except those on treatment IND for approved indications).
* Other anti-Kaposi's sarcoma/HIV drugs.
* Corticosteroids (other than topical).
* Biologic response modifiers.
* Megestrol acetate.
* Agents known to cause neutropenia.
* Trimethoprim/sulfamethoxazole in excess of 160 mg trimethoprim and 800 mg sulfamethoxazole thrice weekly.
* Cytotoxic chemotherapy.

Concurrent Treatment:

Excluded:

* Radiation therapy including electron beam irradiation (other than limited electron-beam radiation to non-marker lesions for treatment of Kaposi's sarcoma).

Patients with the following prior conditions are excluded:

* Prior history of significant cardiac disease or anomaly.
* History of agranulocytosis or severe grade 3 drug-induced neutropenia or documented abnormalities in granulocyte function.

Prior Medication:

Excluded:

* AZT within 14 days prior to study entry.
* Acyclovir as prophylaxis for herpes within 48 hours prior to study entry.

Excluded within 30 days prior to study entry:

* Interferon.
* Biologic response modifiers.
* Cytotoxic chemotherapy.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Blood or cellular blood product. Active illicit drug abuse (specifically cocaine, amyl nitrate, heroin, or other cardioactive agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA School of Medicine, Los Angeles, California
  - Northwestern Univ Med School, Chicago, Illinois

REFERENCES:
- [Background] Petit RG, Miles S, Magpantay L, Mitsuyasu R. Vesnarinone inhibits AIDS-KS cells in culture. Int Conf AIDS. 1994 Aug 7-12;10(1):169 (abstract no PB0104)